CLINICAL TRIAL: NCT05027022
Title: Lower Body and Lower Extremity Flexibility and Strength do Not Correlate With Standing, Stooping and Crouching Performances
Brief Title: Lower Body and Extremity Flexibility and Strength do Not Correlate With Standing, Stooping and Crouching Performances
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, UMUT ERASLAN, PhD, Pamukkale University
Other Study IDs: 601167887/85229
Record Dates: First submitted 2021-08-25; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Flexibility; Strength
Keywords: flexibility, musclestrength, standing, stooping, crouching

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Standing, stooping and crouching are considered important physical demands of the work, which are among the 20 physical work demands defined in the Dictionary of Occupational Titles(1, 2). Agricultural workers, underground miners, aircraft baggage handlers, plumbers, mechanics and many other workers adopt these postures(3-7). These postures are also used in daily activities such as gardening, shopping andcleaning(8).Standing describes an upright position without moving(2). Maintaining this position requires sustained musclea ctivity in various muscles of the body known as the antigravity muscles(9). Stooping consists of bending the torso forward and down with the legs in a relatively straight position. Crouching is an activity performed with the flexion of the hip, knee and ankle while the trunk is in a vertical position. During stooping, the lower back and posterior leg muscles are stretched. Crouching involves similar length changes, particularly in the quadriceps and ankle plantar flexor muscles, as a result of significant flexion in the knee and ankle joints.Unlike standing, as the hip and knee joints are fully flexed during crouching, activation of the quadriceps and calf muscles is potentially required to support lower extremities and weight transfer between limbs(10).

Consideration of the flexibility defined as the maximum range of motion, and the muscular strength associated with the amount of external force a muscle can exert(11, 12), may provide a different perspective to the health care professionals during the interpretation of the work or daily activities. Knowing the relationship between standing, stooping and crouching performances with the direct measurement methods such as flexibility and strength may help to make a more accurate decision during the health care assessments and guiding individuals who have difficulties in these activities to the appropriate rehabilitation program. Starting from this point of view, in this study, we aimed to evaluate the relationship between flexibility and muscular strength tests with standing, stooping and crouching performances.

DETAILED DESCRIPTION:
Participants Over the age of 18, 97 sedentary young adults studying at university were included in this cross-sectional study by convenience sampling. Announcement about the study was made via e-mail and social media.Individuals who volunteered to participate in the study and met the inclusion criteria were enrolled.Inclusion criteria were the absence of any orthopaedic, neurological, rheumatologic or metabolic diseases that cause musculoskeletal involvement, and the absence of a history of surgery on the related extremities. Individuals who had acquired the skills to practice these tests before the study and who had regular physical activity or sports participation (exercising at least 150 minutes per week) were excluded from the study (13). The research protocol was approved by the Institutional Review Board. Written informed consent was obtained from all participants before the study.

Assessments After questioning the demographic characteristics of the volunteers, modified sit-and-reach (MSR), isometric back-leg strength (IBLS) and Valpar 9 Whole Body Range of Motion (WBROM)tests were completed with the participants who met the eligibility criteria. After detailed explanation, the tests were applied to the participants under the supervision of the same physiotherapistin the school of physiotherapy. Firstly WBROM, then IBLS and MSR tests were performed. After each test, participants were given a rest period of 10 minutes in a sitting position.

To evaluate standing, stooping and crouching performances, WBROM test was used.This testprovides information on range of motion, agility and endurance.In this test, which took approximately 30 minutes, the participant was positioned in front of the test panel with the upper frame 6 inches above the head. The participant unscrewed the 22 nuts to release and transfer three different shapes in the standing position in the first transfer, in the standing and stooping positions in the second, in the stooping and crouching positions in the third and in the crouching and standing positions in the last transfer, and retightened the nuts to fix the shapes. This test assesses participants' ability to stand, stoop and crouchwhile performing a manual task. The completion time of each transfer and total time were recorded as seconds(Christopherson & Hayes, 2006; Dailey, Keffala, & Sluka, 2015; Schult, Söderback, & Jacobs, 1995).

MSR test was performed using Baseline™ modified sit and reach box with adjustable measuring bar. It has been reported in the literature that the standard SR test does not take into account differences in limb lengths or proportional differences between legs and arms, which is an important limitation of the test. MSR test that eliminates the possibility of error by creating a relative zero point for each case has been developed due to potential errors that may arise from differences in limb-length ratio between individuals (Hoeger, Hopkins, Button, & Palmer, 1990). At the beginning of this test, while the head, back and hips were against the wall and the soles of the feet were against the block, hands were placed on top of each other and the arms were extended to the front. In this position, only scapular abduction was performed while the head and back were in contact with the wall. The point where the fingertip touches the sliding measuring apparatus was determined as the individual relative zero point. After the determination of the initial position, the SR test was performed as standard. The participant was asked to reach out slowly with hands on top of each other and to advance the movable part of the test device with fingertips. The mean value of three trials was recorded in centimeters (cm).

Isometric back and leg muscle strengths were assessed using a Baseline dynamometer. The dynamometer was connected via a hook to a platform with an adjustable chain. For isometric leg muscle strength assessment, participants were asked to spread their feet at shoulder width on the dynamometer platform and hold the dynamometer bars in forearm pronation position with both hands. After the participant was positioned with the knees slightly flexed, the head and back straight and the projection of the hip joint passing through the ankle, isometric leg strength was evaluated by asking the participant to extend the knees with maximum force vertically. A similar procedure was used for back muscle strength assessment. For this test, the participants were positioned with knees extended, trunk slightly flexed, arms straight and palms facing themselves. In this position, isometric back strength was evaluated by asking the participant to do back extension with maximum force. Leg and back muscle strength measurements were performed three times with one minute pause after each measurement and the mean value in kilograms (kg) was recorded (Hu et al., 2007).

Statistical analysis The data obtained from the participants were recorded in SPSS 18.0 statistical analysis program. Mean and standard deviation were calculated for descriptive data determined by measurement, and number and percentage (%) values were presented for descriptive data determined by counting. Since parametric conditions were met, Pearson Correlation Analysis was used to analyze the relationship between flexibility and muscular strength with standing, stooping and crouching performances. Significance level was accepted as p <0.05.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria were the absence of any orthopaedic, neurological, rheumatologic or metabolic diseases that cause musculoskeletal involvement, and the absence of a history of surgery on the related extremities. healthy young adults who were between 18-35 years old were included.

Exclusion Criteria: Individuals who had acquired the skills to practice these tests before the study and who had regular physical activity or sports participation (exercising at least 150 minutes per week) were excluded from the study. Participants who didn't want to involve this study was excluded.

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Over the age of 18, 97 sedentary young adults studying at university
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
work performances | 30 minutes
  WBROM test was used.This testprovides information on range of motion, agility and endurance.In this test, which took approximately 30 minutes, the participant was positioned in front of the test panel with the upper frame 6 inches above the head. The participant unscrewed the 22 nuts to release and transfer three different shapes in the standing position in the first transfer, in the standing and stooping positions in the second, in the stooping and crouching positions in the third and in the crouching and standing positions in the last transfer, and retightened the nuts to fix the shapes. The completion time of each transfer and total time were recorded as seconds.
flexibility | 10 minutes
  MSR test was performed using Baseline™ modified sit and reach box with adjustable measuring bar.At the beginning of this test, while the head, back and hips were against the wall and the soles of the feet were against the block, hands were placed on top of each other and the arms were extended to the front. In this position, only scapular abduction was performed while the head and back were in contact with the wall. The point where the fingertip touches the sliding measuring apparatus was determined as the individual relative zero point. The participant was asked to reach out slowly with hands on top of each other and to advance the movable part of the test device with fingertips. The mean value of three trials was recorded in centimeters (cm).
strength | 10 minutes
  Isometric back and leg muscle strengths were assessed using a Baseline dynamometer. For this test, the participants were positioned with knees extended, trunk slightly flexed, arms straight and palms facing themselves. In this position, isometric back strength was evaluated by asking the participant to do back extension with maximum force. Leg and back muscle strength measurements were performed three times with one minute pause after each measurement and the mean value in kilograms (kg) was recorded

CONTACTS AND LOCATIONS:
Overall Officials: umut eraslan, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)